CLINICAL TRIAL: NCT01995513
Title: A PHASE 4, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY OF CONTINUED ENZALUTAMIDE TREATMENT BEYOND PROGRESSION IN PATIENTS WITH CHEMOTHERAPY-NAÏVE METASTATIC CASTRATION-RESISTANT PROSTATE CANCER
Brief Title: Safety Study of Continued Enzalutamide Treatment In Prostate Cancer Patients
Acronym: PLATO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDV3100-10; 2013-000722-54 (EudraCT Number); C3431013 (Other: Alias Study Number); PLATO, C3431013 (Other: Alias Study Number)
Record Dates: First submitted 2013-11-18; First posted 2013-11-26 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; abiraterone; Abiraterone Acetate; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enzalutamide & Abiraterone/prednisone (Experimental): Enzalutamide (160 mg) administered as four 40-mg capsules by mouth once daily in combination with abiraterone (1000 mg) administered as four 250-mg tablets by mouth once daily and prednisone (10 mg) administered as one 5-mg tablet by mouth twice daily
  Interventions: Drug: Enzalutamide; Drug: Abiraterone; Drug: Prednisone
- Enzalutamide placebo & Abiraterone/prednisone (Active Comparator): Enzalutamide placebo (placebo) capsules (identical in appearance to enzalutamide) administered as 4 capsules by mouth once daily in combination with abiraterone (1000 mg) administered as four 250-mg tablets by mouth once daily and prednisone (10 mg) administered as one 5-mg tablet by mouth twice daily.
  Interventions: Drug: Abiraterone; Drug: Placebo for Enzalutamide; Drug: Prednisone

INTERVENTIONS:
Drug: Enzalutamide — 160 mg by mouth once daily
  Other Names: MDV3100; Xtandi
  Arms: Enzalutamide & Abiraterone/prednisone
Drug: Abiraterone — 1000 mg by mouth once daily
  Other Names: Abiraterone acetate; Zytiga
Drug: Placebo for Enzalutamide — Sugar pill manufactured to mimic Enzalutamide 40 mg capsule
  Arms: Enzalutamide placebo & Abiraterone/prednisone
Drug: Prednisone — 5 mg by mouth twice daily
  Other Names: prednisolone

SUMMARY:
The purpose of this study is to determine if continued treatment with Enzalutamide is effective in patients with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men with metastatic castration-resistant prostate cancer
* Progressive disease on androgen deprivation therapy
* Patients must agree to continue androgen deprivation therapy with a GnRH agonist/antagonist throughout the study or have had a prior bilateral orchiectomy
* ECOG performance score ≤ 1
* Estimated life expectancy of ≥ 12 months

Exclusion Criteria:

* Prior cytotoxic chemotherapy, aminoglutethimide, ketoconazole, abiraterone, or enzalutamide for the treatment of prostate cancer
* Prior participation in a clinical trial of an investigational agent that inhibits the androgen receptor or androgen synthesis (unless the treatment was placebo)
* History of brain metastasis, active leptomeningeal disease or seizure
* Severe cardiovascular or hepatic disease
* Pituitary or adrenal dysfunction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 509 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Medical Director, Study Director — Medviation, Inc.
Locations (93):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - eResearch Technology, Philadelphia, Pennsylvania
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
- Australia (35):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Ramsay Health Care Australia Pty Ltd, Albury, New South Wales
  - Regional Imaging Border, Albury, New South Wales
  - Terry White Chemist, Albury, New South Wales
  - Concord Cancer Centre, Medical Oncology Department, Concord, New South Wales
  - Concord Hospital Clinical Trials Pharmacy, Concord, New South Wales
  - Epic Pharmacy Lismore, Lismore, New South Wales
  - Macquarie University Hospital Pharmacy, North Ryde, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Epic Pharmacy Port Macquarie base hospital, Port Macquarie, New South Wales
  - Port Macquarie Base Hospital,North Coast Cancer Institute, Port Macquarie, New South Wales
  - North Shore Radiology and Nuclear Medicine, St Leonards, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Sydney Adventist Hospital, Sydney, New South Wales
  - Northern NSW Local Health District, Tweed Heads, New South Wales
  - Queensland Diagnostic Imaging, Tweed Heads, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Regional Imaging, West Albury, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - River City Pharmacy - APHS, Auchenflower, Queensland
  - Icon Cancer Care Chermside, Chermside, Queensland
  - Gold Coast Radiology PTY LTD, Hope Island, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Icon Cancer Care, South Brisbane, Queensland
  - South Coast Radiology, Tugun, Queensland
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Cancer Care SA Pty Ltd, Kurralta Park, South Australia
  - Tenpharm Pty Ltd trading as EPIC Pharmacy Tennyson, Kurralta Park, South Australia
  - Moorabbin Radiology, Bentleigh East, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Cabrini Health - Cabrini Hospital, Malvern, Victoria
  - Border Medical Oncology, Wodonga, Victoria
- Belgium (3):
  - Algemeen Ziekenhuis Groeninge, Kortrijk, West-vlaanderen
  - Cliniques universitaires saint-Luc, Brussels
  - Universitaire Ziekenhuizen Leuven, Leuven
- Denmark (4):
  - Rigshospitalet CPC 7521, Copenhagen, Norrebro
  - Arhus Universitetshospital, Arhus N
  - Rigshospitalet, Copenhagen
  - Frederiksberg Hospital, Frederiksberg
- Finland (3):
  - Helsingin yliopistollinen keskussairaala, Meilahden sairaala, Helsinki
  - Oulun yliopistollinen sairaala, Oulu
  - Tampereen yliopistollinen Sairaala, Tampere
- Institut Gustave Roussy - Service d'Urologie, Villejuif, France
- Italy (11):
  - U.O. Oncologia Medica, IRCCS Istituto Scientifico Romagnolo per lo Studio e la Cura, Meldola, FC
  - Medicina Nucleare, Azienda Ospedaliera "Istituti Ospitalieri" di Cremona, Cremona
  - Servizio di Radiologia, Azienda Ospedaliera "Istituti Ospitalieri" di Cremona, Cremona
  - Struttura Complessa di Oncologia, Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - Laboratorio Farmaci Antiblastici, Meldola (FC)
  - UO Radiologia, Meldola (FC)
  - SCDU Oncologia Medica II Pad, A.O.U. San Luigi Gonzaga, Orbassano to
  - SCDU Radiodiagnostica, A.O.U. San Luigi Gonzaga, Orbassano to
  - SS Medicina Nucleare, A.O.U. San Luigi Gonzaga, Orbassano to
  - Azienda Ospedaliera S. Camillo Forlanini, UOC per il governo clinico in Oncologia Medica, Roma
  - UOC Radiologia Piasta, Azienda Ospedaliera S. Camillo Forlanini, Roma
- Slovakia (9):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Institut nuklearnej a molekularnej mediciny, Banská Bystrica
  - Bratislavske radiodiagnosticke centrum,a.s., Bratislava
  - CUIMED, s.r.o., urologicka ambulancia, Bratislava
  - Univerzitna nemocnica martin, Martin
  - Jessenius-diagnosticke centrum, a.s., Nitra
  - Uroexam, spol. s r.o., Urologicka ambulancia, Nitra
  - IZOTOPCENTRUM, s.r.o., Nitra
  - GAMMALAB, spol.s r.o., Oddelenie nuklearnej mediciny, Trnava
- Spain (9):
  - Hospital Universitario Son Espases, Palma, Balearic Islands
  - CO Badalona-Instituto Germans Trias i Pujol, Badalona, Barcelona
  - ICO Badalona-Instituto Germans Trias i Pujol, Badalona, Barcelona
  - ALTAHIA, Xarxa Assistencial Universitaria de Manresa, Manresa, Barcelona
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona
  - ICO Badalona-Instituto Germans Trias i Pujol, Badalona, Barcelon
  - Hospital del Mar, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Madrid Sanchinarro, Madrid
- Sweden (6):
  - Urologmottagningen, Gothenburg
  - Urologiska kliniken, Malmo
  - Oriola, Mölnlycke
  - Apoteket AB Kliniska Provningar Molnlycke, Mölnlycke
  - Rontgenkliniken, Örebro
  - Urologmottagningen, Örebro
- United Kingdom (7):
  - East and North Hertfordshire NHS Trust, Northwood, Middlesex
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Velindre NHS Trust, Cardiff
  - University College Hospitals NHS Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Oxford University Hospitals NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Attard G, Borre M, Gurney H, Loriot Y, Andresen-Daniil C, Kalleda R, Pham T, Taplin ME; PLATO collaborators. Abiraterone Alone or in Combination With Enzalutamide in Metastatic Castration-Resistant Prostate Cancer With Rising Prostate-Specific Antigen During Enzalutamide Treatment. J Clin Oncol. 2018 Sep 1;36(25):2639-2646. doi: 10.1200/JCO.2018.77.9827. Epub 2018 Jul 20. PMID 30028657

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received enzalutamide in first open label treatment period. Participants in second open label treatment period could cross over to receive abiraterone and prednisone. In double blind period participants were randomized to receive treatment with enzalutamide or placebo, each in combination with abiraterone and prednisone.
Groups:
- Enzalutamide 160 mg: Participants who only received enzalutamide 160 mg as four 40 mg capsules, orally once daily until disease progression (as defined by radiographic imaging or unequivocal clinical progression or death on study), intolerable toxicity, or participant withdrawal, whichever occurred first. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first.
- Enzalutamide 160 mg Crossing Over to Abiraterone 1000 mg+ Prednisone 10 mg: Participants who received (after switching from enzalutamide), in second open label period, abiraterone 1000 mg as four 250 mg tablets, orally once daily and prednisone 10 mg administered as two 5 mg tablets, orally twice daily until disease progression (as defined by radiographic imaging or unequivocal clinical progression or death on study), intolerable toxicity, or participant withdrawal, whichever occurred first. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first.
- Enzalutamide 160 mg+ Abiraterone 1000 mg+ Prednisone 10mg: Participants with confirmed prostate-specific antigen (PSA) progression at Week 21 in open label period, received enzalutamide 160 mg as four 40 mg capsules, orally once daily along with abiraterone 1000 mg as four 250-mg tablets, orally once daily and prednisone 5 mg tablet, orally twice daily in double blind treatment period, up to disease progression (as defined by radiographic imaging or unequivocal clinical progression or death on study), intolerable toxicity, or participant withdrawal, whichever occurred first. Participants were followed up for 16 weeks at a 4-week interval after discontinuation of study drug for survival and subsequent antineoplastic therapy for prostate cancer.
- Placebo + Abiraterone 1000 mg+ Prednisone 10 mg: Participants with confirmed PSA progression at Week 21 in open label period, received placebo matched to enzalutamide as four 40 mg capsules, orally once daily along with abiraterone 1000 mg as four 250-mg tablets, orally once daily and prednisone 5 mg tablet, orally twice daily in double blind treatment period, up to disease progression (as defined by radiographic imaging or unequivocal clinical progression or death on study), intolerable toxicity, or participant withdrawal, whichever occurred first. Participants were followed up for 16 weeks at a 4-week interval after discontinuation of study drug for survival and subsequent antineoplastic therapy for prostate cancer.
Period: Period 1: First Open Label Treatment
Arm/Group | Enzalutamide 160 mg | Enzalutamide 160 mg Crossing Over to Abiraterone 1000 mg+ Prednisone 10 mg | Enzalutamide 160 mg+ Abiraterone 1000 mg+ Prednisone 10mg | Placebo + Abiraterone 1000 mg+ Prednisone 10 mg
Started | 509 | 0 | 0 | 0
Completed | 264 | 0 | 0 | 0
Not Completed | 245 | 0 | 0 | 0
Not completed — Other | 34 | 0 | 0 | 0
Not completed — Death | 14 | 0 | 0 | 0
Not completed — Adverse Event | 40 | 0 | 0 | 0
Not completed — Failure to Achieve PSA response at Week 13 | 43 | 0 | 0 | 0
Not completed — Disease Progression | 92 | 0 | 0 | 0
Not completed — Protocol Non-Compliance | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 20 | 0 | 0 | 0
Period: Period 1: Second Open Label Treatment
Arm/Group | Enzalutamide 160 mg | Enzalutamide 160 mg Crossing Over to Abiraterone 1000 mg+ Prednisone 10 mg | Enzalutamide 160 mg+ Abiraterone 1000 mg+ Prednisone 10mg | Placebo + Abiraterone 1000 mg+ Prednisone 10 mg
Started | 0 | 13 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 13 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 0
Not completed — Disease Progression | 0 | 11 | 0 | 0
Period: Period 2: Double Blind Treatment
Arm/Group | Enzalutamide 160 mg | Enzalutamide 160 mg Crossing Over to Abiraterone 1000 mg+ Prednisone 10 mg | Enzalutamide 160 mg+ Abiraterone 1000 mg+ Prednisone 10mg | Placebo + Abiraterone 1000 mg+ Prednisone 10 mg
Started | 0 | 0 | 126 | 125
Treated | 0 | 0 | 125 | 124
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 126 | 125
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 3 | 3
Not completed — Disease Progression | 0 | 0 | 104 | 107
Not completed — Adverse Event | 0 | 0 | 14 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 5 | 8
Not completed — Protocol Non-Compliance | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT (Intent to treat) population included all participants randomly assigned to study treatment.
Groups:
- Enzalutamide 160 mg: Participants received enzalutamide 160 mg as four 40 mg capsules, orally once daily until disease progression (as defined by radiographic imaging or unequivocal clinical progression or death on study), intolerable toxicity, or participant withdrawal, whichever occurred first. Participants were followed-up until 30 days after last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first.
Arm/Group | Enzalutamide 160 mg
Number analyzed (Participants) | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (8.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 509

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS = time from randomization to first documentation of radiographic progression (RP),unequivocal clinical progression or death due to any cause (death within 112 days of treatment discontinuation without objective evidence of RP),whichever occurred first as per investigator. Unequivocal disease progression was pain requiring chronic administration of analgesics, decline of prostate cancer of Eastern Cooperative Oncology Group (ECOG) performance status score to 3 or higher or initiation of new anticancer therapy/radiation therapy or surgical intervention due to tumor progression. ECOG score range= 0(no severity) to 5(maximum severity).RP for bone disease was evaluated by appearance of 2 or more new bone lesions as per Prostate Cancer Clinical Trials Working Group 2 (PCWG2) or for soft tissue disease according to Response Evaluation Criteria in Solid Tumor version 1.1. Participants with no PFS event at analysis date were censored at last tumor assessment date prior to data cutoff date.
Time Frame: From randomization until disease progression, last tumor assessment without disease progression or death due to any cause, whichever occurred first (maximum up to 20.3 months)
Population: ITT population included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg: Participants with confirmed PSA progression at Week 21 in open label period, received enzalutamide 160 mg as four 40 mg capsules, orally once daily along with abiraterone 1000 mg as four 250-mg tablets, orally once daily and prednisone 5 mg tablet, orally twice daily in double blind treatment period, up to disease progression (as defined by radiographic imaging or unequivocal clinical progression or death on study), intolerable toxicity, or participant withdrawal, whichever occurred first. Participants were followed up for 16 weeks at 4-week interval after discontinuation of study drug for survival and subsequent antineoplastic therapy for prostate cancer.
- Placebo+Abiraterone 1000mg+ Prednisone 10mg: Participants with confirmed PSA progression at Week 21 in open label period, received placebo matched to enzalutamide as four 40 mg capsules, orally once daily along with abiraterone 1000 mg as four 250-mg tablets, orally once daily and prednisone 5 mg tablet, orally twice daily in double blind treatment period, up to disease progression (as defined by radiographic imaging or unequivocal clinical progression or death on study), intolerable toxicity, or participant withdrawal, whichever occurred first. Participants were followed up for 16 weeks at 4-week interval after discontinuation of study drug for survival and subsequent antineoplastic therapy for prostate cancer.
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 126 | 125
months | 5.7 [4.6 to 8.1] | 5.6 [4.5 to 7.3]
Statistical Analysis 1: Comparison: Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg vs Placebo+Abiraterone 1000mg+ Prednisone 10mg; Test type: Superiority or Other; p = 0.2176, Log Rank — P-value was based on log-rank test stratified by PSA response (greater than or equal to [>=] 0 percent [%] to less than [<] 30% vs >=30%) at Week 13 in the open-label period; Hazard Ratio (HR) = 0.828, 95% CI 2-sided [0.612 to 1.119] — Hazard ratio was based on a Cox regression model (with treatment as the only covariate) stratified by PSA response (>=0% to <30% vs >=30%) at Week 13 in the open-label period and is relative to Enzalutamide-placebo with < 1 favoring Enzalutamide

2. Secondary Outcome: Time to Prostate Specific Antigen (PSA) Progression
Description: Time from date of randomization to the date of first confirmed PSA progression as per Prostate Cancer Clinical Trials Working Group 2 (PCWG2). For participant's whose PSA decreased at Week 13 after randomization, progression was defined as 25 percent (%) PSA increase relative to nadir or absolute increase of >=2 nanogram/milliliter (ng/mL) above nadir. Progression was confirmed if another assessment measured at least 3 weeks later met the criterion as well. For participant's whose PSA did not decrease at Week 13 after randomization, progression was defined as 25% PSA increase relative to baseline assessed 12 weeks after baseline. Participants who were not known to have had a PFS event at the analysis date were censored at last PSA assessment date prior to data cutoff date.
Time Frame: From randomization until disease progression, last tumor assessment without disease progression, whichever occurred first (maximum up to 11.1 months)
Population: ITT population included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 126 | 125
months | 2.8 [2.8 to 2.9] | 2.8 [2.8 to 2.8]
Statistical Analysis 1: Comparison: Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg vs Placebo+Abiraterone 1000mg+ Prednisone 10mg; Test type: Superiority or Other; p = 0.4500, Log Rank — P-value was based on log-rank test stratified by PSA response (>=0% to <30% vs >=30%) at Week 13 in the open-label period; Hazard Ratio (HR) = 0.874, 95% CI 2-sided [0.617 to 1.239] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Prostate Specific Antigen (PSA) Response Rate
Description: PSA response rate was defined as percentage of participants with >=30% and >=50% decrease in PSA from baseline at randomization to the maximal PSA response with a threshold of 30% and 50% respectively. PSA response was confirmed if another assessment measured at least 3 weeks later met the criterion as well.
Time Frame: as for outcome 2
Population: Evaluable ITT population included all participants with a PSA value at baseline of Period 2 and at least 1 post baseline assessment. Here, N signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 124 | 122
percentage of participants
  >= 50% | 0.8 [0.0 to 4.4] | 2.5 [0.5 to 7.0]
  >= 30% | 2.4 [0.5 to 6.9] | 2.5 [0.5 to 7.0]
Statistical Analysis 1: Comparison: Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg vs Placebo+Abiraterone 1000mg+ Prednisone 10mg; This analysis is reported for participants with >=50% decrease from baseline in PSA response; Test type: Superiority or Other; p = 0.3101, Cochran-Mantel-Haenszel — P-value was based on Cochran-Mantel-Haenszel mean score test stratified by PSA response (>=0% to <30% vs >=30%) at Week 13 in the open-label period; Difference in Response Rate = -1.65, 95% CI 2-sided [-4.82 to 1.51] — Difference in response rate was based upon standard normal approximation
Statistical Analysis 2: Comparison: Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg vs Placebo+Abiraterone 1000mg+ Prednisone 10mg; This analysis is reported for participants with >=30% decrease from baseline in PSA response; Test type: Superiority or Other; p = 0.9917, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Response Rate = -0.04, 95% CI 2-sided [-3.90 to 3.82] — Difference in response rate was based upon standard normal approximation

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate as assessed by the investigator according to Response Evaluation Criteria in Solid Tumor version 1.1 (RECIST v1.1) was defined as 1) Percentage of participants with confirmed best overall complete response (CR) and partial response (PR); 2) Percentage of participants with CR, PR and stable disease (SD) for target lesions or non-progressive disease for non-target lesions. CR: Disappearance of all non-nodal target and non-target lesions, including target and non-target lymph nodes reduction to <10 millimeter (mm) in short axis. No new lesions and disappearance of all non-target lesions. PR: >= 30% decrease in sum of diameters of target lesions, compared to the sum at baseline. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions.
Time Frame: From randomization until CR or PR, whichever occurred first (maximum up to 21.3 months)
Population: ITT population (with measurable disease at screening) included all participants randomly assigned to study treatment. Here, N signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 38 | 40
percentage of participants
  CR + PR | 0.0 [0.00 to 9.25] | 5.0 [0.61 to 16.92]
  CR + PR + SD | 68.4 [51.35 to 82.50] | 57.5 [40.89 to 72.96]
Statistical Analysis 1: Comparison: Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg vs Placebo+Abiraterone 1000mg+ Prednisone 10mg; This analysis is reported for participants with CR+PR; Test type: Superiority or Other; p = 0.1653, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Objective Response Rate = -5.00, 95% CI 2-sided [-11.75 to 1.75] — Difference in objective response rate was based upon standard normal approximation
Statistical Analysis 2: Comparison: Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg vs Placebo+Abiraterone 1000mg+ Prednisone 10mg; This analysis is reported for participants with CR+PR+SD; Test type: Superiority or Other; p = 0.3216, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Objective Response Rate = 10.92, 95% CI 2-sided [-10.37 to 32.21] — Difference in objective response rate was based upon standard normal approximation

5. Secondary Outcome: Rate of Pain Progression
Description: Rate of pain progression was defined as percentage of participants with an increase of >=30% from baseline in the mean Brief Pain Inventory-Short Form (BPI-SF) pain intensity item scores of 4 items assessing average, worst, least, and intermediate pain severity. BPI-SF is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. BPI-sf includes 4 questions that assess pain intensity (worst, least, average, right now) and 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). BPI-sf score range for each item was from 0=no pain to 10=worst possible pain. Total score was reported as average of individual questions ranges from 0 to 10, where lower scores indicated less pain or less pain interference.
Time Frame: Month 6
Population: ITT population included all participants randomly assigned to study treatment. Here, N signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 58 | 59
percentage of participants | 36.2 [24.0 to 49.9] | 27.1 [16.4 to 40.3]
Statistical Analysis 1: Comparison: Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg vs Placebo+Abiraterone 1000mg+ Prednisone 10mg; Test type: Superiority or Other; p = 0.2963, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Progression Rate = 9.09, 95% CI 2-sided [-7.69 to 25.87] — Difference in Progression Rate was based upon normal approximation

6. Secondary Outcome: Time to First Use of New Antineoplastic Therapy for Prostate Cancer
Description: It was defined as time from randomization to the date of first use of subsequent antineoplastic therapy for prostate cancer. For participants who had not started subsequent antineoplastic therapy as of data analysis cutoff date, the time to first use of subsequent antineoplastic therapy was censored at the date of last assessment.
Time Frame: From randomization until date of first use of any antineoplastic therapy (after last dose date of Period 2, maximum up to 22.3 months
Population: ITT population included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 126 | 125
months | 10.3 [8.7 to 12.1] | 8.6 [7.4 to 11.7]
Statistical Analysis 1: Comparison: Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg vs Placebo+Abiraterone 1000mg+ Prednisone 10mg; Test type: Superiority or Other; p = 0.3818, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.861, 95% CI 2-sided [0.616 to 1.204] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by Functional Assessment of Cancer Therapy-Prostate (FACT-P) Global Score
Description: The FACT-P is a multidimensional, self-reported quality of life instrument consisting of 27 core items that assess participant function in 4 domains: physical, social/family, emotional, functional well-being, and supplemented by 12 site-specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert-type scale, and then combined to produce subscale scores for each domain, as well as a global quality of life score which is the sum of all 5 domain scores and ranges from 0 to 156 where higher scores represent better quality of life.
Time Frame: Baseline, Week 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73, 77, 81, 85, 89
Population: ITT population included all participants randomly assigned to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 126 | 125
units on a scale
  Baseline: number analyzed (Participants) | 125 | 123
  Baseline | 116.4 (20.10) | 119.0 (19.08)
  Change at Week 9: number analyzed (Participants) | 102 | 105
  Change at Week 9 | -3.3 (14.90) | -2.2 (13.90)
  Change at Week 13: number analyzed (Participants) | 88 | 87
  Change at Week 13 | -4.4 (14.44) | -0.5 (13.02)
  Change at Week 17: number analyzed (Participants) | 83 | 77
  Change at Week 17 | -3.7 (12.40) | -2.3 (13.90)
  Change at Week 21: number analyzed (Participants) | 69 | 65
  Change at Week 21 | -2.5 (12.33) | -2.7 (13.57)
  Change at Week 25: number analyzed (Participants) | 61 | 61
  Change at Week 25 | -3.1 (13.47) | -2.1 (10.87)
  Change at Week 29: number analyzed (Participants) | 51 | 49
  Change at Week 29 | -6.8 (13.98) | 0.3 (12.10)
  Change at Week 33: number analyzed (Participants) | 44 | 43
  Change at Week 33 | -5.9 (15.35) | -0.2 (12.90)
  Change at Week 37: number analyzed (Participants) | 35 | 33
  Change at Week 37 | -6.1 (14.25) | 0.9 (12.57)
  Change at Week 41: number analyzed (Participants) | 31 | 29
  Change at Week 41 | -5.7 (12.17) | 1.3 (14.13)
  Change at Week 45: number analyzed (Participants) | 28 | 26
  Change at Week 45 | -6.0 (9.56) | -2.6 (16.27)
  Change at Week 49: number analyzed (Participants) | 27 | 18
  Change at Week 49 | -4.2 (11.36) | 1.8 (10.74)
  Change at Week 53: number analyzed (Participants) | 20 | 15
  Change at Week 53 | -4.8 (10.17) | 1.8 (14.68)
  Change at Week 57 (n =17, 13): number analyzed (Participants) | 17 | 13
  Change at Week 57 (n =17, 13) | -4.3 (9.73) | 0.1 (7.45)
  Change at Week 61: number analyzed (Participants) | 13 | 10
  Change at Week 61 | -5.5 (10.63) | 0.6 (12.94)
  Change at Week 65: number analyzed (Participants) | 13 | 7
  Change at Week 65 | -7.0 (7.86) | 1.9 (9.50)
  Change at Week 69: number analyzed (Participants) | 10 | 7
  Change at Week 69 | -3.5 (11.37) | 4.4 (13.29)
  Change at Week 73: number analyzed (Participants) | 8 | 1
  Change at Week 73 | -0.7 (7.26) | -35.0 (NA) — As only 1 participant was analyzed at Week 73, standard deviation could not be calculated.
  Change at Week 77: number analyzed (Participants) | 7 | 2
  Change at Week 77 | -4.0 (9.81) | 6.5 (30.41)
  Change at Week 81: number analyzed (Participants) | 2 | 0
  Change at Week 81 | 10.8 (9.24) |
  Change at Week 85: number analyzed (Participants) | 2 | 0
  Change at Week 85 | -5.5 (3.54) |
  Change at Week 89: number analyzed (Participants) | 1 | 0
  Change at Week 89 | -2.0 (NA) — As only participant was analyzed at Week 89, standard deviation could not be calculated. |

8. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by Functional Assessment of Cancer Therapy-Prostate (FACT-P) Social/Family Well-Being Domain Scores
Description: The FACT-P is a multidimensional, self-reported quality of life instrument consisting of 27 core items that assess participant function in 4 domains: physical, social/family, emotional, functional well-being, and supplemented by 12 site-specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert-type scale, and then combined to produce subscale scores for each domain. Total subscale score range for social/family well-being domain is from 0 (worst response) to 32 (best response), where higher score indicate better quality of life.
Time Frame: Baseline, Week 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73, 77, 81, 85, 89
Population: ITT population included all participants randomly assigned to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 126 | 125
units on a scale
  Baseline: number analyzed (Participants) | 125 | 123
  Baseline | 22.1 (5.80) | 22.4 (4.84)
  Change at Week 9: number analyzed (Participants) | 104 | 108
  Change at Week 9 | -0.5 (4.33) | -0.8 (4.13)
  Change at Week 13: number analyzed (Participants) | 89 | 89
  Change at Week 13 | -0.4 (3.46) | -0.4 (3.86)
  Change at Week 17: number analyzed (Participants) | 84 | 80
  Change at Week 17 | -0.1 (3.68) | -0.6 (4.64)
  Change at Week 21: number analyzed (Participants) | 70 | 67
  Change at Week 21 | -0.5 (3.24) | -1.2 (5.75)
  Change at Week 25: number analyzed (Participants) | 62 | 62
  Change at Week 25 | 0.1 (2.79) | -1.0 (5.25)
  Change at Week 29: number analyzed (Participants) | 51 | 50
  Change at Week 29 | -0.1 (3.20) | -0.2 (5.18)
  Change at Week 33: number analyzed (Participants) | 44 | 44
  Change at Week 33 | -0.2 (3.21) | 0.0 (4.95)
  Change at Week 37: number analyzed (Participants) | 36 | 33
  Change at Week 37 | -0.8 (3.04) | 0.8 (2.79)
  Change at Week 41: number analyzed (Participants) | 31 | 29
  Change at Week 41 | -1.4 (3.75) | -0.1 (3.51)
  Change at Week 45: number analyzed (Participants) | 28 | 27
  Change at Week 45 | -0.9 (3.36) | -0.8 (3.75)
  Change at Week 49: number analyzed (Participants) | 27 | 18
  Change at Week 49 | -0.6 (2.88) | 0.0 (2.65)
  Change at Week 53: number analyzed (Participants) | 21 | 15
  Change at Week 53 | -1.0 (3.15) | 0.4 (2.56)
  Change at Week 57: number analyzed (Participants) | 17 | 13
  Change at Week 57 | -2.0 (3.06) | 0.2 (1.29)
  Change at Week 61: number analyzed (Participants) | 13 | 10
  Change at Week 61 | -1.5 (2.77) | -0.2 (1.80)
  Change at Week 65: number analyzed (Participants) | 13 | 7
  Change at Week 65 | -1.5 (2.54) | -0.5 (0.96)
  Change at Week 69: number analyzed (Participants) | 10 | 7
  Change at Week 69 | -1.4 (2.03) | -0.5 (0.96)
  Change at Week 73: number analyzed (Participants) | 8 | 1
  Change at Week 73 | -0.6 (3.22) | -1.0 (NA) — As only 1 participant was analyzed at Week 73, standard deviation could not be calculated.
  Change at Week 77: number analyzed (Participants) | 7 | 2
  Change at Week 77 | -0.9 (3.41) | -0.5 (0.71)
  Change at Week 81: number analyzed (Participants) | 2 | 0
  Change at Week 81 | 6.2 (5.42) |
  Change at Week 85: number analyzed (Participants) | 2 | 0
  Change at Week 85 | -1.0 (1.41) |
  Change at Week 89: number analyzed (Participants) | 1 | 0
  Change at Week 89 | 0.0 (NA) — As only 1 participant was analyzed at Week 89, standard deviation could not be calculated. |

9. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by Functional Assessment of Cancer Therapy-Prostate (FACT-P) Emotional Well-Being Domain Scores
Description: The FACT-P is a multidimensional, self-reported quality of life instrument consisting of 27 core items that assess participant function in 4 domains: physical, social/family, emotional, functional well-being, and supplemented by 12 site-specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert-type scale, and then combined to produce subscale scores for each domain. Total subscale score range for emotional well-being domain is from 0 (worst response) to 24 (best response), where higher score indicate better quality of life.
Time Frame: Baseline, Week 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73, 77, 81, 85, 89
Population: ITT population included all participants randomly assigned to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 126 | 125
units on a scale
  Baseline: number analyzed (Participants) | 126 | 124
  Baseline | 18.1 (3.80) | 18.5 (4.06)
  Change at Week 9: number analyzed (Participants) | 104 | 107
  Change at Week 9 | -0.1 (2.81) | 0.1 (3.40)
  Change at Week 13: number analyzed (Participants) | 91 | 88
  Change at Week 13 | -0.1 (3.55) | 0.2 (3.09)
  Change at Week 17: number analyzed (Participants) | 84 | 79
  Change at Week 17 | -0.2 (3.44) | 0.4 (2.88)
  Change at Week 21: number analyzed (Participants) | 71 | 67
  Change at Week 21 | 0.3 (3.48) | 0.1 (3.36)
  Change at Week 25: number analyzed (Participants) | 62 | 63
  Change at Week 25 | 0.3 (2.58) | 0.3 (3.33)
  Change at Week 29: number analyzed (Participants) | 51 | 51
  Change at Week 29 | -0.5 (3.56) | 0.3 (3.27)
  Change at Week 33: number analyzed (Participants) | 44 | 45
  Change at Week 33 | 0.1 (3.33) | 0.9 (2.99)
  Change at Week 37: number analyzed (Participants) | 36 | 34
  Change at Week 37 | -0.7 (4.04) | 0.9 (2.49)
  Change at Week 41: number analyzed (Participants) | 31 | 30
  Change at Week 41 | 0.1 (2.99) | 1.4 (2.60)
  Change at Week 45: number analyzed (Participants) | 28 | 27
  Change at Week 45 | -0.5 (3.23) | 1.2 (2.76)
  Change at Week 49: number analyzed (Participants) | 27 | 19
  Change at Week 49 | 0.0 (3.00) | 1.3 (2.75)
  Change at Week 53: number analyzed (Participants) | 21 | 16
  Change at Week 53 | 0.1 (2.72) | 1.2 (3.23)
  Change at Week 57: number analyzed (Participants) | 17 | 14
  Change at Week 57 | -0.4 (2.32) | 1.6 (2.53)
  Change at Week 61: number analyzed (Participants) | 13 | 11
  Change at Week 61 | -0.3 (3.14) | 1.1 (3.62)
  Change at Week 65: number analyzed (Participants) | 13 | 7
  Change at Week 65 | -0.9 (3.57) | 2.9 (2.54)
  Change at Week 69: number analyzed (Participants) | 10 | 8
  Change at Week 69 | -0.5 (2.93) | 1.5 (2.93)
  Change at Week 73: number analyzed (Participants) | 8 | 2
  Change at Week 73 | 1.0 (2.83) | -5.0 (5.66)
  Change at Week 77: number analyzed (Participants) | 7 | 2
  Change at Week 77 | 0.1 (2.67) | 2.0 (2.83)
  Change at Week 81: number analyzed (Participants) | 2 | 0
  Change at Week 81 | 1.5 (3.54) |
  Change at Week 85: number analyzed (Participants) | 2 | 0
  Change at Week 85 | -1.5 (0.71) |
  Change at Week 89: number analyzed (Participants) | 1 | 0
  Change at Week 89 | -3.0 (NA) — As only 1 participant was analyzed at Week 89, standard deviation could not be calculated. |

10. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by Functional Assessment of Cancer Therapy-Prostate (FACT-P) Functional Well-Being Domain Scores
Description: The FACT-P is a multidimensional, self-reported quality of life instrument consisting of 27 core items that assess participant function in 4 domains: physical, social/family, emotional, functional well-being, and supplemented by 12 site-specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert-type scale, and then combined to produce subscale scores for each domain. Total subscale score range for functional well-being domain is from 0 (worst response) to 28 (best response), where higher score indicate better quality of life.
Time Frame: Baseline, Week 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73, 77, 81, 85, 89
Population: ITT population included all participants randomly assigned to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 126 | 125
units on a scale
  Baseline: number analyzed (Participants) | 126 | 124
  Baseline | 20.2 (5.54) | 20.3 (5.84)
  Change at Week 9: number analyzed (Participants) | 104 | 107
  Change at Week 9 | -1.0 (4.23) | -0.7 (4.62)
  Change at Week 13: number analyzed (Participants) | 91 | 87
  Change at Week 13 | -1.2 (4.07) | -0.4 (4.54)
  Change at Week 17: number analyzed (Participants) | 84 | 78
  Change at Week 17 | -1.3 (4.00) | -0.5 (4.11)
  Change at Week 21: number analyzed (Participants) | 71 | 67
  Change at Week 21 | -1.2 (5.03) | -0.7 (4.03)
  Change at Week 25: number analyzed (Participants) | 62 | 63
  Change at Week 25 | -1.0 (3.41) | -0.3 (4.41)
  Change at Week 29: number analyzed (Participants) | 51 | 51
  Change at Week 29 | -2.4 (4.67) | -0.2 (4.38)
  Change at Week 33: number analyzed (Participants) | 44 | 44
  Change at Week 33 | -2.0 (5.14) | -0.7 (4.49)
  Change at Week 37: number analyzed (Participants) | 36 | 44
  Change at Week 37 | -1.5 (5.22) | 0.2 (5.72)
  Change at Week 41: number analyzed (Participants) | 31 | 30
  Change at Week 41 | -2.1 (4.44) | 0.8 (5.74)
  Change at Week 45: number analyzed (Participants) | 28 | 28
  Change at Week 45 | -2.0 (3.37) | -0.3 (6.28)
  Change at Week 49: number analyzed (Participants) | 27 | 19
  Change at Week 49 | -2.1 (4.55) | 1.5 (5.02)
  Change at Week 53: number analyzed (Participants) | 21 | 16
  Change at Week 53 | -1.6 (4.67) | 1.3 (4.92)
  Change at Week 57: number analyzed (Participants) | 17 | 14
  Change at Week 57 | -1.4 (4.06) | 2.0 (4.37)
  Change at Week 61: number analyzed (Participants) | 13 | 11
  Change at Week 61 | -0.8 (3.34) | 2.9 (5.56)
  Change at Week 65: number analyzed (Participants) | 13 | 7
  Change at Week 65 | -1.2 (2.21) | 1.7 (2.75)
  Change at Week 69: number analyzed (Participants) | 10 | 8
  Change at Week 69 | 0.2 (1.48) | 2.3 (4.23)
  Change at Week 73: number analyzed (Participants) | 8 | 2
  Change at Week 73 | -0.6 (3.02) | 4.0 (12.73)
  Change at Week 77: number analyzed (Participants) | 7 | 2
  Change at Week 77 | -1.6 (3.91) | 2.5 (9.19)
  Change at Week 81: number analyzed (Participants) | 2 | 0
  Change at Week 81 | -1.5 (7.78) |
  Change at Week 85: number analyzed (Participants) | 2 | 0
  Change at Week 85 | -1.5 (2.12) |
  Change at Week 89: number analyzed (Participants) | 1 | 0
  Change at Week 89 | 1.0 (NA) — As only 1 participant was analyzed at Week 89, standard deviation could not be calculated. |

11. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by Functional Assessment of Cancer Therapy-Prostate (FACT-P) Prostate Cancer Domain Scores
Description: The FACT-P is a multidimensional, self-reported quality of life instrument consisting of 27 core items that assess participant function in 4 domains: physical, social/family, emotional, functional well-being, and supplemented by 12 site-specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert-type scale, and then combined to produce subscale scores for each domain. Total subscale score range for prostate cancer domain is from 0 (worst response) to 48 (best response), where higher score indicated better quality of life with fewer symptoms.
Time Frame: Baseline, Week 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73, 77, 81, 85, 89
Population: ITT population included all participants randomly assigned to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 126 | 125
units on a scale
  Baseline: number analyzed (Participants) | 126 | 124
  Baseline | 33.2 (6.85) | 34.2 (6.45)
  Change at Week 9: number analyzed (Participants) | 104 | 107
  Change at Week 9 | -0.7 (5.97) | -0.9 (5.18)
  Change at Week 13: number analyzed (Participants) | 90 | 89
  Change at Week 13 | -1.9 (5.91) | -0.1 (5.36)
  Change at Week 17: number analyzed (Participants) | 84 | 79
  Change at Week 17 | -1.0 (5.36) | -1.4 (5.10)
  Change at Week 21: number analyzed (Participants) | 71 | 67
  Change at Week 21 | -0.4 (5.13) | -0.6 (4.83)
  Change at Week 25: number analyzed (Participants) | 61 | 63
  Change at Week 25 | -0.8 (6.93) | -0.8 (4.42)
  Change at Week 29: number analyzed (Participants) | 52 | 51
  Change at Week 29 | -1.3 (5.75) | -0.3 (4.77)
  Change at Week 33: number analyzed (Participants) | 44 | 45
  Change at Week 33 | -1.4 (5.16) | -0.6 (4.88)
  Change at Week 37: number analyzed (Participants) | 35 | 34
  Change at Week 37 | -1.5 (4.88) | -0.8 (4.32)
  Change at Week 41: number analyzed (Participants) | 31 | 30
  Change at Week 41 | -1.0 (5.13) | -0.7 (5.34)
  Change at Week 45: number analyzed (Participants) | 28 | 28
  Change at Week 45 | -0.8 (4.88) | -1.7 (7.02)
  Change at Week 49: number analyzed (Participants) | 27 | 19
  Change at Week 49 | -0.8 (4.26) | -0.9 (4.63)
  Change at Week 53: number analyzed (Participants) | 20 | 16
  Change at Week 53 | -1.1 (3.65) | -1.8 (5.78)
  Change at Week 57: number analyzed (Participants) | 17 | 14
  Change at Week 57 | -0.5 (3.67) | -3.3 (4.48)
  Change at Week 61: number analyzed (Participants) | 13 | 11
  Change at Week 61 | -2.1 (4.29) | -3.1 (5.68)
  Change at Week 65: number analyzed (Participants) | 13 | 7
  Change at Week 65 | -2.0 (4.05) | -2.6 (6.32)
  Change at Week 69: number analyzed (Participants) | 10 | 8
  Change at Week 69 | -1.5 (3.30) | 1.1 (5.79)
  Change at Week 73: number analyzed (Participants) | 8 | 2
  Change at Week 73 | -0.2 (3.17) | -6.4 (9.32)
  Change at Week 77: number analyzed (Participants) | 7 | 2
  Change at Week 77 | -1.0 (3.71) | -1.5 (13.44)
  Change at Week 81: number analyzed (Participants) | 2 | 0
  Change at Week 81 | 3.1 (1.22) |
  Change at Week 85: number analyzed (Participants) | 2 | 0
  Change at Week 85 | -0.5 (0.71) |
  Change at Week 89: number analyzed (Participants) | 1 | 0
  Change at Week 89 | 0.0 (NA) — As only 1 participant was analyzed at Week 89, standard deviation could not be calculated. |

12. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by Functional Assessment of Cancer Therapy-Prostate (FACT-P) Physical Well-Being Domain Scores
Description: The FACT-P is a multidimensional, self-reported quality of life instrument consisting of 27 core items that assess participant function in 4 domains: physical, social/family, emotional, functional well-being, and supplemented by 12 site-specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert-type scale, and then combined to produce subscale scores for each domain. Total subscale score range for physical well-being domain is from 0 (worst response) to 28 (best response), where higher score indicate better quality of life.
Time Frame: Baseline, Week 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73, 77, 81, 85, 89
Population: ITT population included all participants randomly assigned to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 126 | 125
units on a scale
  Baseline: number analyzed (Participants) | 126 | 124
  Baseline | 22.9 (4.50) | 23.6 (4.42)
  Change at Week 9: number analyzed (Participants) | 105 | 109
  Change at Week 9 | -0.8 (4.04) | 0.1 (3.20)
  Change at Week 13: number analyzed (Participants) | 91 | 89
  Change at Week 13 | -1.0 (4.11) | 0.0 (2.63)
  Change at Week 17: number analyzed (Participants) | 85 | 80
  Change at Week 17 | -1.1 (3.26) | -0.3 (2.97)
  Change at Week 21: number analyzed (Participants) | 70 | 68
  Change at Week 21 | -0.8 (3.11) | -0.8 (4.48)
  Change at Week 25: number analyzed (Participants) | 62 | 63
  Change at Week 25 | -1.7 (4.23) | -0.4 (2.90)
  Change at Week 29: number analyzed (Participants) | 51 | 51
  Change at Week 29 | -2.5 (4.89) | 0.3 (2.67)
  Change at Week 33: number analyzed (Participants) | 44 | 45
  Change at Week 33 | -2.5 (5.37) | 0.1 (3.18)
  Change at Week 37: number analyzed (Participants) | 36 | 34
  Change at Week 37 | -1.8 (4.50) | 0.4 (3.13)
  Change at Week 41: number analyzed (Participants) | 31 | 30
  Change at Week 41 | -1.5 (3.94) | 0.4 (2.80)
  Change at Week 45: number analyzed (Participants) | 28 | 28
  Change at Week 45 | -2.0 (3.72) | -0.4 (3.59)
  Change at Week 49: number analyzed (Participants) | 27 | 19
  Change at Week 49 | -0.9 (3.78) | 0.6 (2.12)
  Change at Week 53: number analyzed (Participants) | 21 | 16
  Change at Week 53 | -0.2 (3.78) | 0.7 (2.85)
  Change at Week 57: number analyzed (Participants) | 17 | 14
  Change at Week 57 | -0.4 (3.25) | 0.4 (2.37)
  Change at Week 61: number analyzed (Participants) | 13 | 11
  Change at Week 61 | -0.8 (3.11) | 0.4 (2.32)
  Change at Week 65: number analyzed (Participants) | 13 | 7
  Change at Week 65 | -1.9 (4.25) | 0.4 (1.99)
  Change at Week 69: number analyzed (Participants) | 10 | 8
  Change at Week 69 | -0.3 (4.08) | -0.5 (2.67)
  Change at Week 73: number analyzed (Participants) | 8 | 2
  Change at Week 73 | -0.3 (2.05) | -3.0 (5.66)
  Change at Week 77: number analyzed (Participants) | 7 | 2
  Change at Week 77 | -0.7 (2.81) | 4.0 (4.24)
  Change at Week 81: number analyzed (Participants) | 2 | 0
  Change at Week 81 | 1.5 (2.12) |
  Change at Week 85: number analyzed (Participants) | 2 | 0
  Change at Week 85 | -1.0 (0.00) |
  Change at Week 89: number analyzed (Participants) | 1 | 0
  Change at Week 89 | 0.0 (NA) — As only 1 participant was analyzed at Week 89, standard deviation could not be calculated. |

13. Secondary Outcome: Time to Degradation of the Functional Assessment of Cancer Therapy-Prostate (FACT-P) Global Score
Description: Time to degradation of FACT-P was defined as the time from randomization to first assessment with at least a 10-point decrease from baseline in the global FACT-P score for each participant. The FACT-P is a multidimensional, self-reported quality of life instrument consisting of 27 core items that assess participant function in 4 domains: physical, social/family, emotional, and functional well-being, and supplemented by 12 site-specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert-type scale, and then combined to produce subscale scores for each domain, as well as a global quality of life score which is the sum of all 5 domain scores and ranges from 0 to 156 with higher scores representing better quality of life. Participants with no score degradation at the time of analysis data cutoff were censored at the date of last assessment showing no degradation.
Time Frame: From randomization up to maximum of 18.4 months
Population: Evaluable ITT population included all participants with a PSA value at baseline of Period 2 and at least 1 post baseline assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 126 | 125
months | 4.6 [3.7 to 6.5] | 6.4 [5.5 to 13.9]
Statistical Analysis 1: Comparison: Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg vs Placebo+Abiraterone 1000mg+ Prednisone 10mg; Test type: Superiority or Other; p = 0.0739, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.399, 95% CI 2-sided [0.967 to 2.025] — [estimate comment as in outcome 1, analysis 1]

14. Other Pre Specified Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment emergent are events between first dose of study drug and up to 30 days after last dose of study drug that were absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious.
Time Frame: Baseline up to 30 days after the last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first (maximum of 99.4 months)
Population: Safety population included all participants who received any amount of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Enzalutamide 160 mg: Participants who only received enzalutamide 160 mg as four 40 mg capsules, orally once daily in the study.
- Enzalutamide Crossing Over to Abiraterone + Prednisone: Participants who received (after switching from enzalutamide) abiraterone 1000 mg as four 250 mg tablets, orally once daily and prednisone 10 mg administered as two 5 mg tablets, orally twice daily in the study.
- Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg: Participants who received enzalutamide 160 mg as four 40 mg capsules, orally once daily along with abiraterone 1000 mg as four 250-mg tablets, orally once daily and prednisone 5 mg tablet, orally twice daily in the study.
- Placebo+Abiraterone 1000mg+ Prednisone 10mg: Participants who received placebo matched to enzalutamide as four 40 mg capsules, orally once daily along with abiraterone 1000 mg as four 250-mg tablets, orally once daily and prednisone 5 mg tablet, orally twice daily in the study.
Arm/Group | Enzalutamide 160 mg | Enzalutamide Crossing Over to Abiraterone + Prednisone | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 509 | 13 | 125 | 124
percentage of participants
  AEs | 93.5 | 100 | 91.2 | 92.7
  SAEs | 32.0 | 30.8 | 37.6 | 29.8

15. Other Pre Specified Outcome: Percentage of Participants With Adverse Events (AEs) Leading to Study Drug Discontinuation
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Outcome of an AE was response to a question answered by the investigator: 'Is the AE leading to study discontinuation or death?' as 'yes'.
Time Frame: as for outcome 14
Population: Safety population included all participants who received any amount of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Enzalutamide Crossing Over to Abiraterone + Prednisone: Participants who received (after switching from enzalutamide), abiraterone 1000 mg as four 250 mg tablets, orally once daily and prednisone 10 mg administered as two 5 mg tablets, orally twice daily in the study.
Arm/Group | Enzalutamide 160 mg | Enzalutamide Crossing Over to Abiraterone + Prednisone | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 509 | 13 | 125 | 124
percentage of participants
  Drug Discontinuation with Enzalutamide or Placebo: number analyzed (Participants) | 509 | 0 | 125 | 124
  Drug Discontinuation with Enzalutamide or Placebo | 11.8 |  | 23.2 | 11.3
  Drug Discontinuation with Abiraterone: number analyzed (Participants) | 0 | 13 | 125 | 124
  Drug Discontinuation with Abiraterone |  | 7.7 | 23.2 | 12.9
  Drug Discontinuation with Prednisone: number analyzed (Participants) | 0 | 13 | 125 | 124
  Drug Discontinuation with Prednisone |  | 7.7 | 16.0 | 12.1

16. Other Pre Specified Outcome: Percentage of Participants With Adverse Events (AEs) Leading to Death
Description: as for outcome 15
Time Frame: as for outcome 14
Population: Safety population included all participants who received any amount of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Enzalutamide Crossing Over to Abiraterone + Prednisone: Participants who received enzalutamide (after switching from enzalutamide), abiraterone 1000 mg as four 250 mg tablets, orally once daily and prednisone 10 mg administered as two 5 mg tablets, orally twice daily in the study.
Arm/Group | Enzalutamide 160 mg | Enzalutamide Crossing Over to Abiraterone + Prednisone | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 509 | 13 | 125 | 124
percentage of participants | 5.9 | 0 | 3.2 | 2.4

17. Other Pre Specified Outcome: Percentage of Participants With Treatment-Emergent Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 30 days after last dose of study drug that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to study drug was assessed by the investigator.
Time Frame: as for outcome 14
Population: Safety population included all participants who received any amount of study drug. "Number Analyzed" signifies participants evaluable for the specified categories for respective arms.
Measure: Number; unit: percentage of participants
Arm/Group | Enzalutamide 160 mg | Enzalutamide Crossing Over to Abiraterone + Prednisone | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo+Abiraterone 1000mg+ Prednisone 10mg
Number analyzed (Participants) | 509 | 13 | 125 | 124
percentage of participants
  TEAEs related to Enzalutamide or Placebo: number analyzed (Participants) | 509 | 0 | 125 | 124
  TEAEs related to Enzalutamide or Placebo | 66.6 |  | 46.4 | 36.3
  TEAEs related to Abiraterone: number analyzed (Participants) | 0 | 13 | 125 | 124
  TEAEs related to Abiraterone |  | 38.5 | 54.4 | 45.2
  TEAEs related to Prednisone: number analyzed (Participants) | 0 | 13 | 125 | 124
  TEAEs related to Prednisone |  | 7.7 | 36.0 | 32.3
  SAEs related to Enzalutamide or Placebo: number analyzed (Participants) | 509 | 0 | 125 | 124
  SAEs related to Enzalutamide or Placebo | 4.1 |  | 7.2 | 4.8
  SAEs related to Abiraterone: number analyzed (Participants) | 0 | 13 | 125 | 124
  SAEs related to Abiraterone |  | 0 | 7.2 | 4.0
  SAEs related to Prednisone: number analyzed (Participants) | 0 | 13 | 125 | 124
  SAEs related to Prednisone |  | 0 | 2.4 | 4.8

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after the last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first (maximum duration of exposure: 99.4 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. The all-cause mortality data was evaluated on all enrolled participants while the data for SAEs and other AEs were evaluated for safety population.
Groups:
- Placebo + Abiraterone 1000 mg + Prednisone 10mg: Participants who received placebo matched to enzalutamide as four 40 mg capsules, orally once daily along with abiraterone 1000 mg as four 250-mg tablets, orally once daily and prednisone 5 mg tablet, orally twice daily in the study.
Arm/Group | Enzalutamide 160 mg | Enzalutamide Crossing Over to Abiraterone + Prednisone | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg | Placebo + Abiraterone 1000 mg + Prednisone 10mg
All-Cause Mortality (participants affected / at risk) | 32/509 | 1/13 | 14/126 | 10/125
Serious Adverse Events (participants affected / at risk) | 163/509 | 4/13 | 47/125 | 37/124
Other Adverse Events (participants affected / at risk) | 474/509 | 13/13 | 113/125 | 113/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide 160 mg (N=509) | Enzalutamide Crossing Over to Abiraterone + Prednisone (N=13) | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg (N=125) | Placebo + Abiraterone 1000 mg + Prednisone 10mg (N=124)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 3 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Exophthalmos (Eye disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 2 | 0 | 0 | 0
Disease progression (General disorders) | 7 | 0 | 2 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 0
General physical health deterioration (General disorders) | 4 | 0 | 1 | 1
Local swelling (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 2 | 0 | 1 | 1
Pyrexia (General disorders) | 3 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0
Abscess jaw (Infections and infestations) | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis tuberculous (Infections and infestations) | 1 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 0 | 1 | 3
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 3 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 6 | 0 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Musculoskeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Dystrophic calcification (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung squamous cell carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3 | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 3 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 3 | 0 | 1 | 0
Nerve root compression (Nervous system disorders) | 2 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 5 | 0 | 5 | 2
Stupor (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 6 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 0 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 2 | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 3 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 11 | 0 | 3 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 3 | 0 | 1 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0 | 2
Ureteric obstruction (Renal and urinary disorders) | 2 | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 2 | 1
Urinary retention (Renal and urinary disorders) | 3 | 0 | 2 | 2
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 2 | 1
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Arterial rupture (Vascular disorders) | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 4 | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide 160 mg (N=509) | Enzalutamide Crossing Over to Abiraterone + Prednisone (N=13) | Enzalutamide 160mg+Abiraterone 1000mg+ Prednisone 10mg (N=125) | Placebo + Abiraterone 1000 mg + Prednisone 10mg (N=124)
Anaemia (Blood and lymphatic system disorders) | 32 | 0 | 5 | 8
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Pernicious anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 4 | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 0 | 3 | 4
Atrial flutter (Cardiac disorders) | 5 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 8 | 1 | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 3 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 1
Chordae tendinae rupture (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 4 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 1 | 1
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 3 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 7 | 0 | 0 | 3
Ventricular extrasystoles (Cardiac disorders) | 4 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 3 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 14 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 2 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1
Cushing's syndrome (Endocrine disorders) | 0 | 1 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 1 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 1 | 0 | 0 | 0
Amaurosis (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 13 | 0 | 2 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 10 | 0 | 2 | 1
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 5 | 0 | 1 | 0
Exophthalmos (Eye disorders) | 2 | 0 | 0 | 1
Eye disorder (Eye disorders) | 1 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 3 | 0 | 0 | 0
Eye pain (Eye disorders) | 2 | 0 | 1 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0
Eyelid margin crusting (Eye disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 2 | 0 | 0 | 0
Iritis (Eye disorders) | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 1 | 0
Macular fibrosis (Eye disorders) | 1 | 0 | 0 | 0
Night blindness (Eye disorders) | 0 | 0 | 1 | 0
Ocular icterus (Eye disorders) | 1 | 0 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 1 | 0 | 0 | 0
Trichiasis (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 3 | 0 | 0 | 3
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 2 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Abasia (General disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 26 | 0 | 5 | 3
Axillary pain (General disorders) | 0 | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 4 | 0 | 2 | 0
Chest pain (General disorders) | 3 | 0 | 5 | 4
Chills (General disorders) | 5 | 0 | 1 | 2
Cyst (General disorders) | 1 | 0 | 0 | 0
Device failure (General disorders) | 2 | 0 | 0 | 1
Device leakage (General disorders) | 0 | 0 | 0 | 1
Device occlusion (General disorders) | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 1
Dysplasia (General disorders) | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 1 | 1
Facial pain (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 206 | 0 | 20 | 19
Feeling abnormal (General disorders) | 4 | 0 | 0 | 0
Feeling drunk (General disorders) | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 8 | 0 | 1 | 2
General physical health deterioration (General disorders) | 5 | 0 | 0 | 0
Hunger (General disorders) | 0 | 0 | 1 | 0
Hyperpyrexia (General disorders) | 1 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 1 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 9 | 0 | 1 | 1
Infusion site extravasation (General disorders) | 1 | 0 | 0 | 1
Injection site swelling (General disorders) | 1 | 0 | 0 | 0
Irritability (General disorders) | 2 | 0 | 1 | 0
Local swelling (General disorders) | 7 | 1 | 6 | 0
Malaise (General disorders) | 5 | 0 | 3 | 0
Medical device complication (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 7 | 0 | 4 | 2
Oedema (General disorders) | 5 | 0 | 3 | 0
Oedema peripheral (General disorders) | 51 | 0 | 8 | 18
Pain (General disorders) | 8 | 0 | 6 | 2
Performance status decreased (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 11 | 0 | 3 | 3
Suprapubic pain (General disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 6 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 8 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 16 | 0 | 7 | 8
Abdominal pain lower (Gastrointestinal disorders) | 4 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 21 | 0 | 0 | 4
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Apical granuloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Breath odour (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 84 | 0 | 22 | 14
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 73 | 0 | 9 | 15
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 0 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 16 | 0 | 5 | 4
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 2 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 12 | 1 | 3 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastric mucosa erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 0 | 4 | 5
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 4 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 3 | 0 | 0 | 2
Large intestine polyp (Gastrointestinal disorders) | 3 | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lip oedema (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 100 | 0 | 23 | 12
Odynophagia (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Oral discharge (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatic disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 2 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 12 | 1 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 29 | 0 | 11 | 2
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 2 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Pneumobilia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1 | 0
Milk allergy (Immune system disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 4 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 0
Atypical mycobacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 5 | 1 | 1 | 2
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 0 | 0 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 1 | 0 | 1 | 0
Cystitis (Infections and infestations) | 5 | 0 | 1 | 2
Diverticulitis (Infections and infestations) | 4 | 0 | 0 | 0
Ear infection (Infections and infestations) | 3 | 0 | 2 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 5 | 0 | 0 | 0
Eyelid infection (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 3 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 2 | 0 | 2 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0
Gastric infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 6 | 0 | 1 | 0
Genital candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Gingival infection (Infections and infestations) | 1 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 2
Helicobacter infection (Infections and infestations) | 1 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 5 | 0 | 5 | 2
Herpes zoster oticus (Infections and infestations) | 1 | 0 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 1 | 0
Infected dermal cyst (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0 | 1
Infection parasitic (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 24 | 1 | 8 | 5
Injection site infection (Infections and infestations) | 1 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Lip infection (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 3 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 20 | 0 | 2 | 4
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Mediastinitis (Infections and infestations) | 1 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 36 | 1 | 0 | 8
Onychomycosis (Infections and infestations) | 3 | 0 | 2 | 1
Oral candidiasis (Infections and infestations) | 9 | 0 | 1 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 2 | 1 | 0 | 0
Otitis media (Infections and infestations) | 2 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 2 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 5 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 5 | 0 | 0 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 5 | 0 | 0 | 3
Skin candida (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 2 | 0
Tooth infection (Infections and infestations) | 5 | 0 | 0 | 2
Tracheitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 30 | 0 | 9 | 5
Urethritis (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 34 | 1 | 10 | 7
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 3 | 0 | 1 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 8 | 0 | 2 | 3
Excoriation (Injury, poisoning and procedural complications) | 5 | 0 | 2 | 2
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 51 | 2 | 14 | 10
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 9 | 0 | 2 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 5 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Periorbital contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 5 | 2 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Skin wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 8 | 6
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 4 | 2
Bacterial test positive (Investigations) | 1 | 0 | 0 | 0
Blood albumin increased (Investigations) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 5 | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 3 | 0 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 2 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 8 | 0 | 3 | 2
Blood glucose increased (Investigations) | 4 | 0 | 1 | 1
Blood iron decreased (Investigations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 1
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 2 | 0 | 2 | 1
Blood pressure orthostatic decreased (Investigations) | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 3 | 0 | 0 | 0
Cardioactive drug level increased (Investigations) | 1 | 0 | 0 | 0
Cystoscopy (Investigations) | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 1
Gamma-glutamyltransferase abnormal (Investigations) | 1 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 6 | 0 | 0 | 2
Heart rate increased (Investigations) | 1 | 0 | 0 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0 | 0
Heart sounds abnormal (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 2 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 3 | 1
Lymph node palpable (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1
Norovirus test positive (Investigations) | 1 | 0 | 0 | 0
Respiratory rate increased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 2 | 0
Troponin increased (Investigations) | 1 | 0 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 1 | 0
Vitamin B12 decreased (Investigations) | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 25 | 0 | 3 | 4
Weight increased (Investigations) | 3 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 83 | 2 | 14 | 11
Dehydration (Metabolism and nutrition disorders) | 5 | 0 | 3 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 1 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 0 | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 0 | 11 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 78 | 2 | 22 | 16
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 112 | 1 | 26 | 28
Bone fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 21 | 1 | 3 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 6 | 0 | 2 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 14 | 1 | 1 | 5
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 2 | 4 | 9
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 21 | 2 | 6 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 27 | 0 | 14 | 7
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 38 | 0 | 13 | 9
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 0 | 2 | 3
Myopathy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 25 | 0 | 2 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 | 1 | 12 | 7
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendon calcification (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 0 | 3 | 1
Benign urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
Choroidal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 1 | 1 | 1 | 0
Amnesia (Nervous system disorders) | 9 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 5 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 8 | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebellar atrophy (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral atrophy (Nervous system disorders) | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 11 | 0 | 2 | 0
Dementia (Nervous system disorders) | 2 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 7 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 49 | 0 | 6 | 5
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 3 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 24 | 0 | 3 | 1
Dyskinesia (Nervous system disorders) | 1 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 50 | 0 | 6 | 3
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Hyperreflexia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 12 | 0 | 5 | 3
Hypoglossal nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Hypokinesia (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 37 | 0 | 3 | 1
Loss of consciousness (Nervous system disorders) | 3 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 16 | 0 | 3 | 2
Migraine (Nervous system disorders) | 3 | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 5 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 23 | 1 | 1 | 0
Parkinson's disease (Nervous system disorders) | 2 | 0 | 0 | 0
Parkinsonian gait (Nervous system disorders) | 1 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0 | 1 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 2 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 4 | 0 | 1 | 1
Radicular pain (Nervous system disorders) | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 10 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 5 | 0 | 0 | 1
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 7 | 0 | 1 | 1
Syncope (Nervous system disorders) | 6 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0
Tongue paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 0 | 0
Tremor (Nervous system disorders) | 5 | 0 | 1 | 3
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 7 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 3 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 16 | 0 | 1 | 2
Apathy (Psychiatric disorders) | 4 | 0 | 0 | 0
Bruxism (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 10 | 0 | 4 | 1
Daydreaming (Psychiatric disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 3 | 0 | 1 | 1
Depressed mood (Psychiatric disorders) | 3 | 0 | 1 | 0
Depression (Psychiatric disorders) | 12 | 1 | 1 | 5
Disorientation (Psychiatric disorders) | 4 | 0 | 0 | 0
Emotional disorder (Psychiatric disorders) | 3 | 0 | 0 | 0
Flat affect (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 2 | 0 | 1 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 40 | 0 | 6 | 6
Mood altered (Psychiatric disorders) | 3 | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 3 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 2 | 0 | 0 | 1
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0
Bladder dysfunction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 2 | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 4 | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 12 | 0 | 1 | 5
Haematuria (Renal and urinary disorders) | 20 | 0 | 6 | 11
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 4 | 0 | 1 | 1
Incontinence (Renal and urinary disorders) | 7 | 0 | 2 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 2 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 7 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 18 | 0 | 1 | 5
Pollakiuria (Renal and urinary disorders) | 13 | 0 | 3 | 4
Polyuria (Renal and urinary disorders) | 1 | 1 | 0 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 2 | 0 | 0 | 1
Strangury (Renal and urinary disorders) | 1 | 0 | 1 | 2
Ureteric obstruction (Renal and urinary disorders) | 3 | 0 | 0 | 0
Urethral dilatation (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urethral pain (Renal and urinary disorders) | 1 | 0 | 2 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urethritis noninfective (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urge incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 18 | 0 | 3 | 2
Urinary retention (Renal and urinary disorders) | 8 | 0 | 2 | 2
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 0 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 3 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 11 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 10 | 0 | 2 | 4
Perineal pain (Reproductive system and breast disorders) | 2 | 0 | 0 | 1
Prostatic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 2 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 1 | 7 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 0 | 6 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 1 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 0
Actinic prurigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 | 0 | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 17 | 0 | 8 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 5 | 0 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0
Solar lentigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Sticky skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 1
Physical assault (Social circumstances) | 1 | 0 | 0 | 0
Cataract operation (Surgical and medical procedures) | 2 | 0 | 0 | 0
Dupuytren's contracture operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Endodontic procedure (Surgical and medical procedures) | 1 | 0 | 0 | 0
Glaucoma surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hip surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0
Mole excision (Surgical and medical procedures) | 1 | 0 | 0 | 0
Nasal polypectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Peripheral nerve decompression (Surgical and medical procedures) | 0 | 0 | 1 | 0
Pterygium operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Skin neoplasm excision (Surgical and medical procedures) | 2 | 0 | 0 | 1
Tendon sheath incision (Surgical and medical procedures) | 1 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 3 | 0 | 0 | 2
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 1 | 1
Flushing (Vascular disorders) | 3 | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 1 | 0
Hot flush (Vascular disorders) | 90 | 1 | 8 | 3
Hypertension (Vascular disorders) | 52 | 0 | 24 | 11
Hypotension (Vascular disorders) | 9 | 0 | 0 | 4
Lymphoedema (Vascular disorders) | 2 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 5 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral coldness (Vascular disorders) | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 3 | 0 | 0 | 0
Phlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.